CLINICAL TRIAL: NCT05912218
Title: REducing Diabetic MacrovascUlar Complications DuE to Peripheral Arterial Disease- REDUCE-PAD
Acronym: REDUCE-PAD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other); Khoo Teck Puat Hospital (Other); National University Health System, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REDUCE-PAD 1
Record Dates: First submitted 2023-05-16; First posted 2023-06-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Peripheral Arterial Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This is a double-blind trial that keeps all patients, study investigators blinded to the treatment. Patients who have met all inclusion criteria and none of the exclusion criteria will be assigned to one of the two study arms (MEDI6570 or normal saline control) in a 1:1 ratio. Randomization will be accomplished using a permuted block scheme with variable block size and will be stratified by study site. The trial will use randomly generated treatment allocations within sealed opaque envelopes. Reconstitution of study drug and normal saline control will be by an unblinded study team member.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEDI6570 (Experimental): Biological MEDI6570,subcutaneous injection
  Interventions: Biological: MEI6570
- Placebo (Placebo Comparator): Saline Control,subcutaneous injection
  Interventions: Biological: MEI6570

INTERVENTIONS:
Biological: MEI6570 — Saline Control
  Other Names: Placebo

SUMMARY:
This is a Phase IIa, multi-centre study conducted at 3 sites in Singapore (SGH and NUHS, KTPH). 70 patients with diabetes mellitus (DM) and peripheral arterial disease (PAD) will be randomised in a ratio 1:1 to receive normal saline control or MEDI6570 400mg by monthly subcutaneous injection for 9 months.

DETAILED DESCRIPTION:
This is a mechanistic, randomised, double-blind, controlled Phase IIa trial that investigates whether 9 months of treatment with MEDI6570 affects lower limb microvascular perfusion and atheroma inflammation and progression. Patients with both DM and PAD will receive monthly subcutaneous injections of 400mg MEDI6570 (in an injection volume of 4.0ml), or injection/volume-matched normal saline control (4.0ml) subcutaneously, every 4 weeks for 32 weeks (9 doses in total). Com

Approximately 70 participants will be randomly assigned to a study intervention, with an anticipated 35 participants being randomized to receive active study intervention, and 35 participants being randomized to receive normal saline control.

The primary objective of the study is to determine whether monthly subcutaneous injections of MEDI6570 for 9 months reduces lower limb atheroma plaque inflammation and improves lower limb microvascular perfusion, when compared to normal saline control.

The primary endpoint in REDUCE-PAD will be the between-group difference (intervention vs. normal saline control) in the change in PET and MRI scan parameters from baseline to 9 months. Efficacy, safety, PK, and immunogenicity of MEDI6570 will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must provide informed consent before any study specific activities are performed, must be able and willing to meet all requirements for randomisation, and must adhere to the schedules of activities.
2. Men must be ≥ 21 years of age at the time of signing the ICF. Women must be ≥ 40 years of age at the time of signing the ICF. For female participants, the participant must not be pregnant or lactating and must be of non-childbearing potential, confirmed at screening Visit 1 by one of the following:

   1. Postmenopausal, defined as amenorrhea for ≥ 12 months following cessation of all exogenous hormonal treatments, and with luteinizing hormone and follicle stimulating hormone levels in the postmenopausal range.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not considered as irreversible surgical sterilization.
3. Participant must have body mass index within the range 18 to 40 kg/m2 inclusive.
4. Participants must have moderate stable PAD (ABI < 0.7 and/or TBI < 0.5) with no prior history of lower limb revascularisation or ulcers.
5. On stable medical therapy for type 2 DM for at least 6 weeks prior to screening with no clinically significant dose change and/or new medications in the recent 6 weeks
6. All male participants should refrain from fathering a child or donating sperm during the study and for 190 days following the last dose. Non-sterilised male study participants should be advised to use a condom for all sexual intercourse with a female partner of childbearing potential from Day 1 through the end of the study follow-up period.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. Uncontrolled Type 1 or Type 2 diabetes defined as haemoglobin A1c (HbA1c) >10%.
3. Increased risk of bleeding

   1. Patients with history or presence of any bleeding disorder.
   2. Signs of ongoing bleeding at screening (e.g., identified macroscopic bleeding, low haemoglobin presumed to be caused by bleeding) or high risk for major bleeding in accordance with the Investigator's assessment.
   3. . Need for chronic therapeutic anticoagulation therapy anticipated to be required throughout the course of the study (short-term treatment with prophylactic doses of heparin/low molecular weight heparin are allowed).
   4. Known severe liver disease (e.g., ascites and/or clinical signs of coagulopathy).
4. History or presence of any of the following:

   1. Cancer within 5 years before randomization, except for non-melanoma skin cancer.
   2. Alcohol or substance abuse within 6 months before randomization, as judged by the investigator.
   3. Known history of hypersensitivity reactions to other biologics, to human IgG preparations, or to any component of MEDI6570, or ongoing severe allergy as judged by the investigator.
   4. Patients with active positive results on screening for serum hepatitis B surface antigen, hepatitis C antibody, or HIV.
5. Any clinically important abnormalities in clinical chemistry, haematology, coagulation parameters, as judged by the investigator, including but not limited to:

   1. AST > 2.0 × ULN.
   2. ALT > 2.0 × ULN.
   3. TBL > 1.5 x ULN (unless due to Gilbert's syndrome).
   4. Platelet count < 100,000 platelets/μl.
6. BP values at screening Visit 1:

   1. Systolic BP < 90 mmHg or > 180 mmHg.
   2. Diastolic BP > 100 mmHg.
   3. Participants who are excluded based on elevated BP may be rescreened following adequate treatment.
7. Any clinically important abnormalities in clinical chemistry, haematology, coagulation parameters, or urinalysis results.
8. History of blood dyscrasia, haemostatic disorder, systemic bleeding, or prior trauma that places the subject at a higher risk of bleeding.
9. Receipt of any investigational device or therapy within 6 months or 5 half-lives before screening (whichever is longer). This criterion does NOT apply for inactive, non-replicating COVID-19 vaccines approved by Health Authorities or under emergency use authorization.
10. Planned participation in an additional investigational study of an intervention or biologic before the end of the follow-up period. Participation in observational studies or studies without investigational drugs or devices is allowed.
11. Participants who are legally institutionalised.
12. An employee or close relative of an employee of the sponsor,

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Lower limb atheroma plaque inflammation | 9 months
  Lower limb atheroma plaque inflammation Changes from baseline to 9 months in lower limb atheroma plaque FDG uptake measured by PET/MRI scans.

SECONDARY OUTCOMES:
Lower limb perfusion | 9 months
  Changes from baseline to 9 months in ankle brachial index (ABI) and toe brachial index (TBI)
Lower limb microvascular perfusion | 9 months
  Changes from baseline to 9 months in lower limb microvascular perfusion measured by MRI scans.
Lower limb atheroma plaque progression | 9 months
  Changes from baseline to 9 months in lower limb atheroma plaque volume measured by US arterial duplex and MRI scans

CONTACTS AND LOCATIONS:
Locations (1):
- Prof Derek J. Hausenloy, Singapore, Singapore, Singapore